CLINICAL TRIAL: NCT01872611
Title: Randomized, Double-Masked, Vehicle Controlled, Clinical Evaluation To Assess The Safety And Efficacy Of Nepafenac Ophthalmic Suspension, 0.3% For Improvement In Clinical Outcomes Among Diabetic Subjects Following Cataract Surgery
Brief Title: Nepafenac Once Daily for Macular Edema - Study 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-12-071; 2013-001874-12 (EudraCT Number)
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Results first posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-06

CONDITIONS: Non-Proliferative Diabetic Retinopathy; Cataract
Keywords: Diabetes Type I; Diabetes Type II; Non-proliferative diabetic retinopathy; Macular edema; Cataract
MeSH Terms: conditions — Cataract; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Macular Edema | interventions — nepafenac; prednisolone acetate; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nepafenac (Experimental): With prednisolone acetate standard of care, Nepafenac Ophthalmic Suspension, 0.3%, 1 drop instilled in the operative eye 1 day prior to surgery, continuing on the day of surgery, and for 90 days following surgery. An additional 1 drop will be administered 30 to 120 minutes prior to surgery.
  Interventions: Drug: Nepafenac Ophthalmic Suspension, 0.3%; Drug: Prednisolone acetate
- Vehicle (Placebo Comparator): With prednisolone acetate standard of care, Nepafenac vehicle, 1 drop instilled in the operative eye 1 day prior to surgery, continuing on the day of surgery, and for 90 days following surgery. An additional 1 drop will be administered 30 to 120 minutes prior to surgery.
  Interventions: Other: Vehicle; Drug: Prednisolone acetate

INTERVENTIONS:
Drug: Nepafenac Ophthalmic Suspension, 0.3%
  Other Names: Test intervention
  Arms: Nepafenac
Other: Vehicle — Inactive ingredients used as placebo comparator
  Other Names: Nepafenac Vehicle
  Arms: Vehicle
Drug: Prednisolone acetate — 1 drop instilled in the operative eye 4 times daily beginning post-operatively on the day of surgery for the first 2 weeks, followed by 2 times daily for the next 2 weeks
  Other Names: Omnipred™; Prednisolone acetate ophthalmic suspension

SUMMARY:
The purpose of this study is to demonstrate superiority of Nepafenac Ophthalmic Suspension, 0.3% dosed once daily relative to Nepafenac Vehicle based upon clinical outcomes among diabetic participants following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Planned cataract extraction by phacoemulsification with implantation of a posterior chamber intraocular lens;
* History of Type 1 or 2 diabetes and non-proliferative diabetic retinopathy (NPDR) (mild, moderate, or severe) in the study eye;
* Best-corrected visual acuity (BCVA) of 73 letters or worse in the study eye with expectation of improvement after surgery;
* Understand and sign an informed consent document;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Pre-existing macular edema in the study eye;
* History in the study eye of retinal detachment, wet age-related macular degeneration, chronic or recurrent inflammatory eye disease, or prior procedures;
* Planned cataract surgery in the fellow eye prior to the Day 90 postoperative study visit or through study exit;
* Planned multiple procedures for the study eye during the cataract/intraocular lens;
* Use of exclusionary medications, including nonsteroidal anti-inflammatory drugs (NSAIDs) and steroids, as specified in protocol.
* Participation in any other clinical study within 30 days of the screening visit;
* Females of childbearing potential who are breast feeding, have a positive urine pregnancy test at screening, are not willing to undergo a urine pregnancy test upon entering or exiting the study, intend to become pregnant during the study, or do not agree to use adequate birth control methods for the duration of the study;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 819 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Lead GCRA, Pharma, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 73 investigational centers located in the U.S., Europe, the Middle East, Africa, Latin America, the Caribbean, and the Asia Pacific region.
Pre-assignment Details: Of the 819 participants enrolled, 191 were exited as screen failures and 23 were discontinued prior to randomization. This reporting group includes all randomized participants (605).
Groups:
- Nepafenac: Nepafenac Ophthalmic Suspension, 0.3%
- Vehicle: Nepafenac Ophthalmic Suspension Vehicle
Period: Overall Study
Arm/Group | Nepafenac | Vehicle
Started | 301 | 304
Randomized | 301 | 304
Treated (Safety Analysis Set) | 293 | 295
Full Analysis Set | 289 | 293
Completed | 277 | 292
Not Completed | 24 | 12
Not completed — Adverse Event | 3 | 1
Not completed — Adverse Event, prior to treatment | 0 | 1
Not completed — Death | 0 | 1
Not completed — Death, prior to treatment | 0 | 1
Not completed — Lost to Follow-up | 8 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Reason not provided | 6 | 6

BASELINE CHARACTERISTICS:
Population: Full analysis set, defined as all randomized participants who completed implant surgery and had at least one on-therapy postsurgical visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nepafenac | Vehicle | Total
Number analyzed (Participants) | 289 | 293 | 582
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (8.5) | 68.1 (8.4) | 67.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 149 | 298
  Male | 140 | 144 | 284

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Best-corrected Visual Acuity (BCVA) Improvement of ≥ 15 Letters From Preoperative Baseline to Day 14 and Maintained Through Day 90
Description: BCVA (with spectacles or other visual corrective devices) was reported in letters read correctly, using the Early Treatment Diabetic Retinopathy Study (ETDRS) test of 70 letters. Improvement of BCVA was defined as an increase (gain) in the number of letters read, compared to the baseline assessment. One eye (study eye) contributed to the analysis.
Time Frame: Baseline to Day 14, and maintained through Day 90
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | Nepafenac | Vehicle
Number analyzed (Participants) | 289 | 293
Percentage of participants | 48.8 | 50.5
Statistical Analysis 1: Comparison: Nepafenac vs Vehicle; This endpoint was considered primary for United States (US) registration and secondary for European Union (EU) registration; Test type: Superiority or Other; p = 0.671, Regression, Logistic; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.7 to 1.3], Standard Error of Mean 0.2 — Parameter dispersion is the standard error for the odds ratio

2. Primary Outcome: Percentage of Participants Who Develop Macular Edema Within 90 Days Following Cataract Surgery (Day 0)
Description: Macular edema was defined as ≥ 30% Increase from pre-operative baseline in central subfield macular thickness, as measured with Spectral Domain Ocular Coherence Tomography (SD-OCT). One eye (study eye) contributed to the analysis.
Time Frame: Day 0 to Day 90
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | Nepafenac | Vehicle
Number analyzed (Participants) | 289 | 293
Percentage of participants | 5.9 | 14.3
Statistical Analysis 1: Comparison: Nepafenac vs Vehicle; This endpoint was considered primary for EU registration and secondary for US registration; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 0.4, 95% CI 2-sided [0.2 to 0.7], Standard Error of Mean 0.1 — Parameter dispersion is the standard error for the odds ratio

3. Secondary Outcome: Percentage of Participants With BCVA Improvement of ≥ 15 Letters From Preoperative Baseline to Day 90
Time Frame: Baseline to Day 90
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | Nepafenac | Vehicle
Number analyzed (Participants) | 289 | 293
Percentage of participants | 65.4 | 65.9

4. Secondary Outcome: Percentage of Participants With BCVA Improvement of ≥ 15 Letters From Preoperative Baseline to Day 60
Time Frame: Baseline to Day 60
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | Nepafenac | Vehicle
Number analyzed (Participants) | 289 | 293
Percentage of participants | 68.9 | 62.1

5. Secondary Outcome: Percentage of Participants With a > 5-letter Loss in BCVA From Day 7 to Any Visit
Time Frame: Day 7 up to any visit through Day 90
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Nepafenac | Vehicle
Number analyzed (Participants) | 289 | 293
percentage of participants | 18.7 | 16.7

6. Secondary Outcome: Percentage of Participants With With a > 10-letter Loss in BCVA From Day 7 to Any Visit
Time Frame: Day 7 up to any visit through Day 90
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Nepafenac | Vehicle
Number analyzed (Participants) | 289 | 293
percentage of participants | 10.7 | 8.9

ADVERSE EVENTS:
Time Frame: Reporting of adverse events (AEs) began once informed consent was obtained and continued through Day 90 (or Day 120, if unresolved macular edema present at Day 90). Ocular adverse events are presented for both study eye and nonstudy eye combined.
Description: An AE was defined as any untoward medical occurrence in a participant after signing the informed consent and did not necessarily have to have a causal relationship with the study treatment. AEs were reported as pretreatment, treatment-emergent, and posttreatment. AEs were obtained through solicited and spontaneous comments from the participants.
Groups:
- Pretreatment: All participants who consented to participate in the study prior to the initiation of study treatment
- Posttreatment: All participants after cessation of study treatment up to study exit
Arm/Group | Pretreatment | Nepafenac | Vehicle | Posttreatment
Serious Adverse Events (participants affected / at risk) | 5/819 | 14/293 | 14/295 | 4/588
Other Adverse Events (participants affected / at risk) | 0/819 | 0/293 | 0/295 | 0/588
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=819) | Nepafenac (N=293) | Vehicle (N=295) | Posttreatment (N=588)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0
Diabetic retinal oedema (Eye disorders) | 0 | 0 | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 0 | 0 | 0 | 1
Posterior capsule rupture (Eye disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Device dislocation (General disorders) | 0 | 1 | 0 | 0
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Arteriovenous fistula operation (Surgical and medical procedures) | 0 | 0 | 1 | 0
Cardiac operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Cataract operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Intra-ocular injection (Surgical and medical procedures) | 0 | 0 | 1 | 0
Skin graft (Surgical and medical procedures) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.